CLINICAL TRIAL: NCT00345488
Title: Fast Track ER Admittance of Hip Fracture Patients
Brief Title: Fast Track Admittance of Hip Fracture Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Other Study IDs: HHSG-DT-01
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2006-06-28 (Estimated); Status verified 2006-05

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The study examines time spent in the emergency room on admission of patients with hip fracture in a cohort with a traditional setup compared with a prospective cohort with a fast track admission schedule including nurse initiation of treatmnet, standardized analgesia, fluid and oxygen therapy and standardized logistics for x-ray and admission procedures.

ELIGIBILITY:
Inclusion Criteria:

* Admission with a primary hip fracture

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2002-09; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD, Principal Investigator — Hvidovre University Hospital